CLINICAL TRIAL: NCT06920199
Title: Clinical Study to Evaluate the Safety and Efficacy of Donor-derived Treg Cell Injection Combined With Recombinant Human Interleukin-2 in the Treatment of Refractory cGVHD Subjects
Brief Title: Treatment of Refractory cGVHD by Donor-derived Treg Cell Injection Combined With Recombinant Human Interleukin-2
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-Treg-cGVHD-2024
Record Dates: First submitted 2025-03-19; First posted 2025-04-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: cGVHD
Keywords: Steroid dependence; Refractory cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: single-arm, open-label, dose-escalation clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor-derived Treg cell injection combined with interleukin 2 (Experimental): Donor-derived Treg cell injection, injections, The first dose was 1.0× 10^6Treg cells /kg, the second dose was 5.0×10^6Treg cells /kg, and the third dose was 10.0×10^6Treg cells /kg,single-dose.
  Interleukin 2,1 million IU/m2/d,last 13 weeks.
  Interventions: Biological: Donor-derived Treg cell injection combined with interleukin 2

INTERVENTIONS:
Biological: Donor-derived Treg cell injection combined with interleukin 2 — Subjects received Treg cell infusion at day D0, and interleukin 2 was administered subcutaneously daily from 1 week before to 12 weeks after infusion.

SUMMARY:
This study is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety, tolerability, changes and persistence of peripheral blood Treg cells, and pharmacodynamic characteristics of donor-derived Treg cell injection combined with recombinant human interleukin-2 in treating subjects with refractory cGVHD，and to preliminarily observe the efficacy of the study drugs in subjects with refractory cGVHD.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety, tolerability, changes and persistence of peripheral blood Treg cells, and pharmacodynamic characteristics of donor-derived Treg cell injection combined with recombinant human interleukin-2 in treating subjects with refractory cGVHD，and to preliminarily observe the efficacy of the study drugs in subjects with refractory cGVHD.In this study, rapid titration of the first dose group and a "3+3" rule design were used for dose escalation to minimize patient exposure to ineffective doses while minimizing the occurrence of risk.Three dose groups were set up: 1×10^6 Treg cells /kg dose group, 5.0×10^6 Treg cells /kg dose group and 10×10^6Treg cells /kg dose group.One infusion per dose group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-70 years old, male or female;
* The subjects had received allo-HSCT, including cord blood transplantation;
* TSubjects with moderate/severe cGVHD that meets the NIH diagnostic criteria (031) for steroid dependence or resistance, meeting one of the following:

  1. There was no improvement in cGVHD in initial treatment patients treated with > 0.5mg/kg/ day or 1 mg/kg/ day every other day for at least 4 weeks;
  2. Steroid dependence: predtisone dose > 0.25 mg/kg/d or > 0.5 mg/kg/qod cGVHD relapse or progression; cGVHD recurred after two attempts to gradually reduce prednisone dose at an interval of at least 8 weeks, with prednisone dose > 0.25 mg/kg/day to be maintained.
* Prednisone dose > 0.25 mg/kg/d for more than 4 weeks; Subjects must maintain a stable prednisone dose for 4 weeks prior to the first Treg cell infusion and not increase or discontinue other immunosuppressants (including cyclosporine, tacrolimus, and sirolimus);
* The ECOG score of the subjects was 0-2;
* the expected survival of the subject is more than 3 months;
* Liver, kidney, heart and lung function meet the following requirements (except liver and kidney dysfunction caused by cGVHD) :

  1. Creatinine clearance (calculated by Cockcroft Gault formula) ≥60 mL/min;
  2. Cardiac ejection fraction greater than 50%, no clinically significant electrocardiogram changes;
  3. Forced expiratory volume (FEV1) in the first second of baseline lung function ≥50%, and FEV1 decline caused by cGVHD could be included;
  4. Total bilirubin ≤2.0ULN; ALT and AST≤3ULN, ALT and AST increases caused by cGVHD could be included in the group.
* Hematopoietic function: neutrophils >1×10^9/L, platelets >25×10^9/L; Supportive treatments such as platelet transfusion and other cytokines are excluded.
* The subject or the subject's guardian can understand this experiment and has signed the informed consent.
* Donor age 14-70 years old, male or female;
* The ECOG score of the donor is 0-1;
* The donor must be a hematopoietic stem cell donor who underwent allo-HSCT prior to the subject;
* Female donors must test negative for serum or urine beta-human chorionic gonadotropin (HCG) within 3 weeks of blood collection;
* The donor can establish the necessary venous access for collection, without the contraindication of white blood cell collection; If peripheral venous leukocyte collection is insufficient, be willing to insert a central catheter; (15) The donor agrees to donate and signs a consent form.

Exclusion Criteria:

* Subjects had a recurrence of primary malignant disease before receiving Treg treatment;
* The subjects had persistent, recurrent or delayed aGVHD;
* Continuous use of prednisone >1 mg/kg/day is required;
* The severity of the subject's cGVHD cannot be assessed by physical examination or laboratory examination;
* overlap syndrome；
* The subjects had major organ (cardio-cerebrovascular, pulmonary) dysfunction not caused by cGVHD, and had previous (within 3 months) gastrointestinal active bleeding; History of uncontrolled hypertension or hypertensive crisis or hypertensive encephalopathy, history or evidence of significant cardiovascular and cerebrovascular risk, including any of the following conditions: congestive heart failure, unstable angina pectoris, clinically significant arrhythmias (e.g., ventricular fibrillation, ventricular tachycardia, etc.); History of arterial thrombosis (such as stroke, transient ischemic attack) within the last 3 months; A history of symptomatic deep vein thrombosis, pulmonary embolism, or coronary angiogenesis, defibrillation, or any clinically relevant complication or disease within the last 6 months that could pose a risk to subject safety or interfere with study evaluation, procedure, or completion;
* The subjects are hemodialysis patients;
* The subject or donor has an active, uncontrolled bacterial, viral, or fungal infection that requires treatment；
* The subjects are pregnant or lactating women; Subjects who plan to become pregnant during the post-transfusion study, or within 1 year of completion or withdrawal from the study;
* Participants who had received IL-2 therapy or drug therapy targeting IL-2 within 4 weeks prior to enrollment；
* Received DLI treatment within 100 days before enrollment;
* Received CAR-T or similar engineered cell therapy within 100 days prior to enrollment;
* Had received new cGVHD therapies (including imatinib, BTK inhibitors, rituximab and other immunosuppressants) within 4 weeks before enrollment after transplantation;
* Have a history of microvascular diseases such as TMA, hemolytic uremic syndrome, thrombotic thrombocytopenic purpura, etc；
* Subjects with poor IL-2 treatment compliance;
* Participants who participated in other CGVHD-related clinical studies within 4 weeks prior to enrollment;
* Subjects who are known to be allergic to any component of Treg cell injection;
* Any situation that the investigator believes would compromise the safety of the subject or interfere with the study purpose, or that the investigator considers it inappropriate to participate in the study;
* Having a medical condition that affects the signing of written informed consent or the inability to follow study procedures; Unwilling or unable to comply with research requirements;
* The donor was a pregnant woman.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of DLT in patients with refractory cGVHD treated with donor-derived Treg cell injection combined with low dose rhIL-2 injection | Up to day 28
  To evaluate the incidence of DLT in patients with refractory cGVHD treated with donor-derived Treg cell injection combined with low dose rhIL-2 injection。
  DLT is defined as any of the following conditions related to the study drug within 28 days after the subject's infusion of Treg cell injection, despite treatment:
  1. Grade 4 or 5 cytokine release syndrome caused by Treg cell injection treatment;
  2. Grade 3 cytokine syndrome caused by Treg cell injection treatment and no remission to grade 2 or below within 7 days;
  3. Occurrence of grade 3 or higher neurotoxicity;
  4. Grade 4 hematologic toxicity: caused by non-underlying disease and lasting ≥ 28 days (except for lymphopenia, neutrophil and thrombocytopenia caused by chemotherapy pretreatment);
  5. Any unanticipated toxicity that necessitates discontinuation of treatment at the discretion of the investigator or collaborating unit.
Incidence of grade 3 and above adverse reactions | Through study completion, an average of 2 year
  Incidence of adverse events associated with the study products；Adverse events assessed according to NCI-CTCAE v5.0.

SECONDARY OUTCOMES:
Evaluate the number of Treg cells in subjects' peripheral blood | An average of 1 year
  Evaluate the number of Treg cells in subjects' peripheral blood after donor-derived Treg cell injection administration
Analysis of the number changes of lymphocyte subsets in peripheral blood. | Through study completion, an average of 2 year
  Analysis of the number changes of lymphocyte subsets in peripheral blood, Including T/B/NK cells.
Score changes in the 36-Item Short Form Health Survey (SF-36) | Through study completion, an average of 2 year
  Adopt 36-Item Short Form Survey (SF-36)to analyze the changes in patients' scores after medication compared with baseline.
Score changes in Lee Chronic Graft-versus-Host Disease Symptom Scale | Through study completion, an average of 2 year
  Adopt 36-Item Short Form Survey (SF-36)to analyze the changes in patients' scores after medication compared with baseline.
Changes in cGVHD severity | Through study completion, an average of 2 year
  Changes in cGVHD severity,according to chronic graft-versus-host disease grading system.
Objective Response Rate (ORR) | Through study completion, an average of 2 year
  To evaluate the efficacy of donor-derived Treg cells combined with low-dose IL-2 in the treatment of refractory cGVHD subjects, including 12 and 24 weeks of ORR.
Patient-reported Outcomes | Through study completion, an average of 2 year
  Reports directly from patients on their own health, functional status, and treatment experience, excluding explanations from health care workers or anyone else. A score of ≥7 on the Lee cGVHD Symptom Scale was associated with improved quality of life.
Proportion of subjects able to reduce steroid requirement to <0.25 mg/kg/ day. | Through study completion, an average of 2 year
  Proportion of subjects able to reduce steroid requirement to <0.25 mg/kg/ day.
Duration of response after administration (DOR) | Through study completion, an average of 2 year
  Duration of response after administration (DOR),Defined as the time between first remission and disease progression, new cGvHD systemic treatment, or all-cause death, whichever occurs first.
Failure-free survival after administration (FFS) | Through study completion, an average of 2 year
  Failure-free survival after administration (FFS),The time from the beginning of cell reinfusion to the first disease progression, recurrence after remission, or death from any cause.
Overall survival | Through study completion, an average of 2 year
  The time from cell retransfusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: xianmin song, Doctor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No